CLINICAL TRIAL: NCT04886466
Title: Importance of Core Stability for Coordinated Movement of the Human Body in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, Ph.D.; senior specjalit of the Rehabilitation Clinc, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/KRN/2019
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: stroke; core stability; muscle tone; motor coordination
MeSH Terms: conditions — Stroke | interventions — Core Stability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The trunk movement coordinated and legs coordination during walking in place. (Experimental): The intervention (active tension of the muscles stabilizing the core) was tested in post-stroke patients (study group).
  Interventions: Procedure: core stability in a sitting position and while walking in one place
- The coordinated movement of the trunk and legs during fast walking in place. (Experimental): The intervention (active tension of the muscles stabilizing the core) was tested in patients with back pain syndrome, but without neurological deficits (control group).
  Interventions: Procedure: core stability in a sitting position and while walking in one place

INTERVENTIONS:
Procedure: core stability in a sitting position and while walking in one place — The intervention consisted of checking how the active tension of the multisection and transverse abdominal muscles affects the pattern of the trunk movement (in the sitting position) and the work of the lower limbs and the speed of movement while walking in a place.

SUMMARY:
This is an observational study. Measurements were made during two different motor tasks: trunk tilts without and with the tension of the abdominal muscles in the sitting position and walking in a place with high knee lifting. It was checked how the intervention (active tension of the muscles stabilizing the core) changes the parameters of the motor coordination of the trunk and lower limbs.

DETAILED DESCRIPTION:
Surface electrodes (single-use 55 and 40 mm; ECG Electrodes; Sorimex, Poland) were glued to the subject's body according to the SENIAM (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles) procedure for the transverse abdominal, multifidus, and supraspinal muscles, and a laser rangefinder was attached to the dorsal side at chest height. Before each exercise, the subject was instructed on how the exercise should be done.

The examination involved two motor exercises. In the first one, the subject was seated on the therapeutic table (with their upper extremities crossed over their chest) and instructed to lean forward as far as possible (ideally to place their torso on their thighs) and then quickly return to their starting position. The movement was repeated three times. Then the subject performed three more repetitions of the movement with their core engaged (i.e., their abdominal muscles contracted or "stabilized"). The range of trunk inclination in the sagittal plane (mm) and in the frontal plane (m), and the reaction of the multifidus, transverse abdominal, and supraspinatus muscles (tension values reported in microvolts [µV]) were measured using a millimeter board, laser pointer, rangefinder (measurement/angle of inclination accuracy of ± 1.5 mm), electrode, and a device for measuring the voltage of selected muscle groups, Luna EMG (accuracy of measurement [-1-+1V+/-1mV]).

The second exercise was a march-in-place with a high elevation of the knees. This exercise was also done as quickly as possible (time measured for 20 steps in place in seconds [s]). The exercise was done in duplicate. On the second occasion, subjects were instructed to do the exercise with their core engaged (i.e., their abdominal muscles contracted or "stabilized"). The exercise was performed in duplicate. The duration of the march and the elevation of the feet were measured, as well as the activity of the multifidus, transverse abdominal, and supraspinatus muscles.

ELIGIBILITY:
Main criteria for stroke group inclusion: 1) patients with ischemic stroke; 2) patients with hemiparesis after 5 to 7 week after stroke; 3) subjects with stable trunk (the Trunk Control Test 70-100 points); 4) subjects who were in a functional state allowing walking (Rankin Scale ≤ 3); 5) no severe deficits in communication, memory, or understanding what can impede proper measurement performance; 6) at least 22 years of age; maximum 83 years of age.

Main criteria for stroke group exclusion: 1) stroke up to five weeks after the episode, 2) epilepsy, 3) lack of trunk stability, 4) lack of independent walking, 5) high or very low blood pressure, dizziness, malaise.

Main criteria for control group inclusion: 1) the control group consisted of subjects with stable trunk (TCT 100 points); correct muscle tension (MAS 0), independent walking; 2) at least 22 years of age; maximum 83 years of age.

Criteria for control group exclusion: 1) a history of neurologic or musculoskeletal disorders such as stroke or brain injury or other conditions that could affect their ability to active movement the trunk and the legs; 2) back pain; 3) no severe deficits in communication, memory, or understanding what can impede proper measurement performance; 4) high or very low blood pressure, dizziness, malaise.

Ages: 22 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Range of active movement of the trunk in frontal plane. | up to 1 week
  The range of trunk inclination in the frontal plane (m) was measured using a millimeter board, laser pointer, rangefinder (measurement/angle of inclination accuracy of ± 1.5 mm).
Range of active movement of the trunk in sagittal plane. | up to 1 week
  The range of trunk inclination in the sagittal plane (mm) was measured using a millimeter board, laser pointer, rangefinder (measurement/angle of inclination accuracy of ± 1.5 mm).
The duration of the march-in-place | up to 1 week
  Time measured for 20 steps using the stopwatch
Elevation of the feet | up to 1 week
  The elevation of the feet were measured using the laser pointer, rangefinder (measurement/angle of inclination accuracy of ± 1.5 mm).
The reaction of the multifidus, transverse abdominal, and supraspinatus muscles. | up to 1 week
  The reaction of muscles (tension values reported in microvolts [µV]) was measured using an electrode, and a device for measuring the voltage of selected muscle groups, Luna EMG (accuracy of measurement [-1-+1V+/-1mV]).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Olczak, PhD, Principal Investigator — Rehabilitation Clinic, Military Institute of Medicine
Locations (1):
- Anna Olczak, Warsaw, Masovian District, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olczak A. Importance of core stability for coordinated movement of the human body in stroke rehabilitation. Neurol Res. 2022 Jan;44(1):7-13. doi: 10.1080/01616412.2021.1950952. Epub 2021 Jul 10. PMID 35040753